CLINICAL TRIAL: NCT03221790
Title: A Study Evaluating the Effects of Low and High FODMAP Diets on Mucosal Protease Nerve Interactions in IBS Patients
Brief Title: Effect of FODMAPs on Mucosal Inflammation in IBS Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Dr. Stephen Vanner, Professor of Medicine, Queen's University
Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 29677
Record Dates: First submitted 2017-06-07; First posted 2017-07-19 (Actual); Last update posted 2017-10-05 (Actual); Status verified 2017-10

CONDITIONS: Irritable Bowel Syndrome With Diarrhea
Keywords: Irritable bowel syndrome; Low FODMAP diet; Mucosal Inflammation
MeSH Terms: conditions — Irritable Bowel Syndrome; Mucositis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Low and High FODMAP Diets in IBS (Experimental): This study will be comprised of the following four time periods: "baseline", "run-in", "low FODMAP diet", and "high FODMAP diet". Participants will undergo baseline assessment with questionnaires on demographics, IBS symptoms (IBS symptom severity scoring questionnaire), diet, and psychological parameters. Baseline mucosal colonic biopsies will be obtained, and metabolome analysis from urine samples. These will be repeated 3 other times during each of the above time periods. Low FODMAP Diet followed by a High FODMAP Diet
  Interventions: Other: Low FODMAP Diet followed by a High FODMAP Diet

INTERVENTIONS:
Other: Low FODMAP Diet followed by a High FODMAP Diet — 3 weeks on a low FODMAP diet followed by 3 weeks on a high FODMAP Diet

SUMMARY:
OBJECTIVE: To gain mechanistic insights, we will compare effects of low fermentable oligosaccharides, disaccharides and monosaccharides and polyols (FODMAP) and high FODMAP diets on symptoms and colonic protease expression in patients with diarrhea predominant irritable bowel syndrome (IBS-D). We will measure how protease changes affect excitability of pain sensing neurons and correlate this with measurements of the metabolome and the microbiome.

DESIGN: We aim to perform a single blind prospective study of patients with diarrhea predominant IBS (Rome IV criteria) who will sequentially consume a high and low FODMAP diets, each for 3 weeks. Symptoms will be assessed using the IBS symptom severity scoring (IBS-SSS). Electrophysiological studies of changes in mouse dorsal root ganglia neurons in response to colonic mucosal/lamina propria supernatants will be carried out. Protease antagonist will be used to specifically assess protease expression. The metabolome will be evaluated using metabolic profiling in urine using mass spectrometry. Stool microbiota composition will be analysed by 16S rRNA gene profiling. All the above testing will be performed at 4 time points: at baseline, 3 weeks following a run-in period, after a 3-week-long high FODMAP diet, and after a 3-week-long low FODMAP diet period.

HYPOTHESIS: We anticipate that colonic tissue protease effects on the excitability of dorsal root ganglia (DRG) neurons will increase with a high FODMAP diet and decrease with a low FODMAP diet, but that this may not be found in all patients. The magnitude of the effect may vary and this variation could be due to differences in the individual patients microbiome.

DETAILED DESCRIPTION:
Up to 15 % of adults in Western society suffer from irritable bowel syndrome (IBS), and it is the second leading cause, behind the common cold, of workplace absenteeism. This proposal addresses critical knowledge gaps in our understanding of IBS mechanisms. What environmental triggers cause pain symptoms to chronically wax and wane? A fundamental observation is that over 70% of IBS patients report that meals trigger abdominal pain and diarrhea. Therefore, we examined the effects of a diet low in fermentable oligo, di, monosaccharides and polyols (FODMAPs) because up to 50-70% IBS patients reported improved symptoms on this diet (McIntosh et al 2016; Halmos et al 2014). We found that symptoms, particularly pain, were markedly improved in IBS patients on a low compared to a high FODMAP diet. Moreover, we found in a subset of patients evidence that FODMAPs activate intestinal mast cells, a major source of proteases and histamine, and their expression appears to be associated with IBS symptoms, although this remains to be proven. Thus, this diet provides a useful clinical tool to stimulate protease activity and study their actions. Sensitization (modulation of intracellular mechanisms leading to exaggerated action potential discharge in response to a given stimulus) of nociceptive dorsal root ganglia (DRG) neurons by tissue mediators is a fundamental mechanism underlying abnormal pain signaling. We also have compelling evidence in human IBS patients that a family of proteases are key mediators underlying another critical knowledge gap that we identified, i.e. which tissue mediators can lead to sustained and amplified abdominal pain. We and others found these proteases are elevated in IBS tissues, and that they sensitize DRG neurons - the primary sensory neurons that innervate the colon. Based on these findings, our goal is to test the overarching hypothesis that diet can trigger recurrent symptoms in IBS through activation of tissue proteases that cause exaggerated pain by signaling to nociceptive DRG neurons. Recurrent exposure to such diet components and the resulting protease signaling is an important cause of the waxing and waning of symptoms over time. Thus, our objective is to characterize the relationship of a specific dietary intervention with protease activity in IBS patients.

This will be a prospective study comparing the effect of low-FODMAP and high-FODMAP on symptoms and protease effects on the excitability of nociceptive DRG neurons. We will analyze the urinary metabolome as a secondary measure of mast cell mediators (i.e. histamine and proteases). We will also collect stool for possible future microbiome analysis as diet microbiome interactions (i.e. fermentation of the FODMAPs) may predict the magnitude of the response. The study will be conducted at Hotel Dieu Hospital's Gastroenterology clinics and endoscopy suite in Kingston, Ontario. This study will be comprised of the following four time periods: "baseline", "run-in", "high FODMAP diet", and "low FODMAP diet". Participants will undergo baseline assessment with questionnaires on demographics, IBS symptoms (IBS symptom severity scoring questionnaire), diet, as well as a questionnaire pertaining to psychological parameters. A detailed questionnaire pertaining to participants' diet will be administered at baseline. Baseline mucosal colonic biopsies will be obtained using limited flexible sigmoidoscopy. Baseline stool microbiota composition will be analysed by 16S rRNA gene profiling. Fecal calprotectin levels will be obtained from stool samples. Urine and blood metabolome will be analysed at baseline also using mass spectrometry. These will be repeated 3 weeks later during a run-in period to assess if these measurements are stable in time or not. This run-in period will be 3 weeks long. After completion of the run-in period, patients will be asked to consume a high FODMAP diet for 3 weeks. All tests carried out at baseline and during the run-in period will be carried out for a third time. Participants will meet with investigators and be given dietary guidance, including a handout outlining foods to eat and avoid. A dietician will be involved extensively in this process to ensure the instructions are adequate and accurate. For the remainder of the study, patients will not be able to take antibiotics, and fibre supplements. After the 3-week-long high FODMAP diet period, participants will meet again with the dietician to obtain instructions on how to consume a low FODMAP diet. After 3 weeks on a low FODMAP diet, all baseline testing will be performed a fourth time. We aim to enroll 20 patients. Based on a 70% response rate to low FODMAP diet (Halmos et al. 2014), and our experience in previous studies, this number should be adequate.

Please note that the biopsies taken at sigmoidoscopy will be processed at HDH for the supernatants, and then frozen for later electrophysiological studies at the Gastro-Intestinal Diseases Research Unit (GIDRU) at KGH.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 18 years of older
* Meet the Rome IV criteria for IBS (abdominal pain or discomfort at least 3 days per month in the last three months associated with two or more of the following: defecation, onset associated with change of frequency of stool or change associated with a change in form of stool. The symptoms must be going on for more than six months and be associated with an absence of routine clinical red flags)

Exclusion Criteria:

* Patients with a history of gastric, small bowel or colonic surgery
* Patients with active Inflammatory Bowel Disease
* Patients with celiac disease
* Patients who are unable or unwilling to come off the following medications: antibiotics, stool bulking agents, narcotics, or lactulose.
* Patients who are already on a low-FODMAP diet or a diet that may be have substantially different FODMAP content from usual Canadian diet (paleolithic diet, specific carbohydrate diet, gluten-free diet, Atkins)
* Patients cannot have used antibiotics in the past 4 weeks.
* Pregnant patients will not be invited to participate. (Sexually active women of child-bearing age will be asked if it is possible that they are pregnant, and if there is a doubt, they will not be invited to participate.) Patients will confirm they are using birth control during the time they are participating in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-11-01 (Estimated); Primary Completion 2018-07-01 (Estimated); Study Completion 2019-02-01 (Estimated)

PRIMARY OUTCOMES:
Change in Rheobase | Colonic Biopsies will be obtained at baseline, 3 weeks later after a run-in period, 3 weeks after a low FODMAP Diet, and 3 weeks after being on a high FODMAP Diet
  Number of IBS patients whose supernatants increased neuronal excitability with high FODMAP vs. Low FODMAP diet ( excitability = rheobase = amount of current needed to elicit a single action potential) measured by patch clamp recording of mouse DRG neurons incubated in response to incubation with proteases in the IBS-D supernatants.

SECONDARY OUTCOMES:
Questionnaires on IBS symptom severity, stool microbiota, urine and blood metabolome | This will be done at baseline, after a 3 week run-in period, after a 3 weeks on a high FODMAP Diet, and after 3 weeks on a low FODMAP Diet
  Number of patients whose symptoms improved with the low FODMAP diets using the IBS-SSS questionnaire
Questionnaire on psychological scores | This will be done at baseline, after a 3 week run-in period, after a 3 weeks on a low FODMAP Diet, and after 3 weeks on a high FODMAP Diet
  The number of patients whose HADS questionnaire worsened with a high FODMAP diet and/or improved with a low FODMAP diet
Stool microbiota analysis | This will be done at baseline, after a 3 week run-in period, after a 3 weeks on a low FODMAP Diet, and after 3 weeks on a high FODMAP Diet
  Number of patients whose 16S RNA profile changed following a low or high FODMAP diet.
Urine Metabolome | This will be done at baseline, after a 3 week run-in period, after a 3 weeks on a high FODMAP Diet, and after 3 weeks on a low FODMAP Diet
  Number of patients whose urine metabolome was altered by a low and high FODMAP diet.
Blood metabolome | This will be done at baseline, after a 3 week run-in period, after a 3 weeks on a high FODMAP Diet, and after 3 weeks on a low FODMAP Diet
  Number of patients whose metabolome in blood was altered by a low and high FODMAP diet.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Vanner, MD, Principal Investigator — Queen's University

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be made available to other researchers

REFERENCES:
- [Background] McIntosh K, Reed DE, Schneider T, Dang F, Keshteli AH, De Palma G, Madsen K, Bercik P, Vanner S. FODMAPs alter symptoms and the metabolome of patients with IBS: a randomised controlled trial. Gut. 2017 Jul;66(7):1241-1251. doi: 10.1136/gutjnl-2015-311339. Epub 2016 Mar 14. PMID 26976734
- [Background] Halmos EP, Power VA, Shepherd SJ, Gibson PR, Muir JG. A diet low in FODMAPs reduces symptoms of irritable bowel syndrome. Gastroenterology. 2014 Jan;146(1):67-75.e5. doi: 10.1053/j.gastro.2013.09.046. Epub 2013 Sep 25. PMID 24076059